CLINICAL TRIAL: NCT00944918
Title: A Partially-blind Phase III Randomised Trial of Fulvestrant (Faslodex) With or Without Concomitant Anastrozole (Arimidex) Compared With Exemestane in Postmenopausal Women With ER+ve Locally Advanced/Metastatic Breast Cancer Following Progression on Non-steroidal Aromatase Inhibitors
Brief Title: Study of Faslodex With or Without Concomitant Arimidex Versus Exemestane Following Progression on Non-steroidal Aromatase Inhibitors (NSAI)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9238UK/0005
Record Dates: First submitted 2009-07-22; First posted 2009-07-23 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Progression-free Survival
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant; Anastrozole; exemestane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): fulvestrant and anastrozole
  Interventions: Drug: fulvestrant; Drug: anastrozole
- 2 (Experimental): fulvestrant and placebo
  Interventions: Drug: fulvestrant
- 3 (Active Comparator): exemestane alone
  Interventions: Drug: exemestane

INTERVENTIONS:
Drug: fulvestrant — Intramuscular injection on days 1, 15, and 29 and then once monthly until disease progression.
  Other Names: Faslodex
  Arms: 1; 2
Drug: anastrozole — Tablet, oral, once daily until disease progression.
  Other Names: Arimidex
  Arms: 1
Drug: exemestane — Tablet, oral, once daily until disease progression.
  Other Names: Aromasin
  Arms: 3

SUMMARY:
A partially-blind, randomised, multicentre phase III trial of Faslodex plus concomitant Arimidex versus Faslodex plus Arimidex-Placebo versus exemestane in postmenopausal locally advanced / metastatic breast cancer patients who have progressed on NSAIs. Randomisation to Faslodex ± Arimidex / Arimidex-Placebo or exemestane will be open (1:1:1). For Faslodex treated patients the randomisation to Arimidex or Arimidex-Placebo will be double-blind.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the breast.
* Metastatic disease must be measurable or evaluable
* Relapsed or progressed during prior treatment with single-agent NSAI, meeting either of the following criteria:
* NSAI given as adjuvant therapy that lasted ≥ 12 months OR
* Achieved an objective CR, PR, or SD that that lasted ≥ 6 months after prior 1st-line
* Female postmenopausal patients

Exclusion Criteria:

* Hormone receptor status1. ER -ve and PgR NK2. ER-ve and PgR -ve3. ER NK
* Prescribed Tamoxifen for metastatic disease
* Rapidly progressive visceral disease
* Patients with malignancies within the last 5 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-12; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 3 months during treatment and, at time of discontinuation from treatment

SECONDARY OUTCOMES:
Objective complete response (CR) and partial response (PR) rate | every 3 months during treatment and, at time of discontinuation from treatment
Duration of response | every 3 months during treatment and, at time of discontinuation from treatment
Clinical benefit (i.e., 6-month CR, PR, and stable disease) rate | every 3 months during treatment and, at time of discontinuation from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Young-Huck Im, Principal Investigator — Professor(Samsung Medical Center)
Locations (2):
- South Korea (2):
  - Research Site, Ilsan
  - Research Site, Seoul

REFERENCES:
- [Derived] Johnston SR, Kilburn LS, Ellis P, Dodwell D, Cameron D, Hayward L, Im YH, Braybrooke JP, Brunt AM, Cheung KL, Jyothirmayi R, Robinson A, Wardley AM, Wheatley D, Howell A, Coombes G, Sergenson N, Sin HJ, Folkerd E, Dowsett M, Bliss JM; SoFEA investigators. Fulvestrant plus anastrozole or placebo versus exemestane alone after progression on non-steroidal aromatase inhibitors in postmenopausal patients with hormone-receptor-positive locally advanced or metastatic breast cancer (SoFEA): a composite, multicentre, phase 3 randomised trial. Lancet Oncol. 2013 Sep;14(10):989-98. doi: 10.1016/S1470-2045(13)70322-X. Epub 2013 Jul 29. PMID 23902874